CLINICAL TRIAL: NCT02377765
Title: A Single Blind, Randomised, Controlled Trial to Evaluate the Effectiveness of Transcutaneous Posterior Tibial Nerve Stimulation (TPTNS) in Overactive Bladder (OAB) Symptoms in Women Responders to Posterior Tibial Nerve Stimulation (PTNS)
Brief Title: Use of Transcutaneous Posterior Tibial Nerve Stimulation (TPTNS) in Maintaining OAB Symptoms Improvement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool Women's NHS Foundation Trust (Other)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LWH0991
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Overactive Bladder
Keywords: Neuromodulation; Detrusor overactivity; Urinary urgency; Urgency urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percutaneus Stimulation (Active Comparator): PTNS performed bilaterally every 4 weeks within the Physiotherapy Department.
  Interventions: Procedure: Percutaneus Stimulation
- Transcutaneous Stimulation (Experimental): TPTNS applied bilaterally, using two surface, self-adhesive, round electrodes (3 cm in diameter) in each leg at least 3 times per week.
  Interventions: Device: Transcutaneous Stimulation

INTERVENTIONS:
Device: Transcutaneous Stimulation — TPTNS through a TENS unit is a non-invasive technique, easily manageable by patients, which lacks some adverse side effects reported with the use of PTNS, such as bleeding and/or pain at the site of needle insertion. As the technique is self-administered, the associated costs might be substantially lower when compared to PTNS, which involves repeated Hospital appointments for maintenance therapy.
  Arms: Transcutaneous Stimulation
Procedure: Percutaneus Stimulation — PTNS aims to stimulate the sacral nerve plexus (origin to the parasympathetic innervations to the bladder) through the afferent fibres of the posterior tibial nerve, a mixed nerve containing L5-S3 fibres (Slovak, Chapple and Barker, 2014). This is achieved by a needle electrode inserted above the medial malleolus. Interestingly, this anatomical area is known as acupuncture point Spleen6 (Sp6).
  Arms: Percutaneus Stimulation

SUMMARY:
This study will help to determine the effectiveness of a self-supervised, home-based Transcutaneous Posterior Tibial Nerve Stimulation treatment protocol in maintaining Overactive Bladder (OAB) symptoms improvement in women responders to Posterior Tibial Nerve Stimulation (PTNS)

DETAILED DESCRIPTION:
Conservative management of OAB includes (NICE, 2006): behavioural therapy (bladder training techniques, prompted voiding, timed voiding…); physical therapy (PFM exercises, Biofeedback, Neuro Muscular Electrical Stimulation…); lifestyle interventions (weight loss, smoking cessation…) and fluid advice (fluid balance, reduction of caffeine intake…). Antimuscarinic agents are recommended if non-pharmacological treatment proves ineffective (NICE, 2006). However, results of behavioural and physical therapy have been shown to fall off by three months after treatment (Burgio et al, 1998). Furthermore, less than one third of patients are compliant with anticholinergic medication after 6 months, mostly due to intolerable side effects, but also to lack of efficacy (Hampel, 2007; Kelleher et al, 1997).

Patients refractory to conservative regimens are candidates in our Physiotherapy Department for peripheral Neuromodulation therapy in the form of Percutaneus Tibial Nerve Stimulation (PTNS). Although its mechanism of action is still poorly understood, its efficacy has been reported to be comparable to that of the antimuscarinic agents, with an objective success rate of 60% (Burton, Sajja & Latthe, 2012), but with a better side effect profile.

TPTNS is a non-invasive technique, easily manageable by patients, which lacks some adverse side effects reported with the use of PTNS, such as bleeding and/or pain at the site of needle insertion. As the technique is self-administered, the associated costs might be substantially lower when compared to PTNS, which involves repeated Hospital appointments for maintenance therapy.

This study will help to determine the effectiveness of a self-supervised, home-based Transcutaneous Posterior Tibial Nerve Stimulation treatment protocol in maintaining Overactive Bladder (OAB) symptoms improvement in women responders to Posterior Tibial Nerve Stimulation (PTNS)

Participants will be assigned to one of the two treatments arms using a computer generated random number table, with assignments drawn from sealed, opaque, serially numbered envelopes.

Participants will be recruited from the Physiotherapy Department at the Liverpool Women's Hospital. Our primary outcome variable will be changes in 24-hour voiding frequency, number of episodes of urgency, as well as number of episodes of urge urinary incontinence. These variables can be reliably measured in self-completed 3-day bladder diaries (Gormley et al, 2012).

As OAB is a symptom-based diagnosis, the quality of life (QoL) impact of the symptoms is a crucial aspect of the condition. We will therefore use as secondary end point the score in the OAB-q questionnaire, a patient-reported outcome measure (PROM) of symptom severity as well as Health Related Quality of Life (HRQOL). The OAB-q has shown good content and construct validity, as well as high internal consistency and good test-retest reliability (Coyne et al, 2006).

Bladder diaries and the OAB-q questionnaire are routinely used in our Department for all patients starting on PTNS (T1). Collection of data will be carried out again at the end of the 12-week course of PTNS. Data obtained at this point (T2) will determine those subjects who are objective responders and who will be invited to enter the trial and be randomized into one of the two treatment arms. During the study period, further assessments will be carried out by the main investigator, who will be blinded to the treatment group allocation, at 6 weeks (T3), 3 months (T4) and 6 months (T5).

PTNS will be performed bilaterally, inserting a 40 mm x 0.25 mm acupuncture needle (Classic Plus Sterile Needle, HMD Europe), three finger breaths cephalad to medial malleolus and posterior to the medial border of the tibia (SP6 acupuncture point). A self-adhesive electrode will be placed on the medial aspect of the calcaneus. The needle and the electrode will be attached to a low voltage electrostimulator (AS SUPER 4 digital, Pierenkemper GmbH, Germany), set up with a pulse duration of 200 μsecs and a frequency of 20 Hz. The amplitude (0-20 mA, adjustable in steps of 0.1 mA) will be increased until flexion of the first toe or fanning of all toes is seen, or tingling sensation in the sole of the foot is reported, always at a tolerable level. Elevation of the Intensity will be allowed whenever the patient describes fading of the above sensation due to accommodation.

TPTNS will be also applied bilaterally, using two surface self-adhesive electrodes in each leg, one placed at SP6 and the other placed on the ankle skin behind the medial malleolus. Electrical stimulation will be applied through a TENS unit (NeuroTrac PelviTone, Verity Medical Ltd, Hampshire, UK) using the same parameters as in the PTNS group.

An experienced Women's Health physiotherapist will conduct the PTNS sessions in the control group and will instruct subjects in the TPTNS group in the stimulation technique. Participants will be provided with a telephone number to contact the research team in case they have any queries or any difficulty with the use of the TENS unit.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Over 18 years of age.
* Clinically diagnosed of idiopathic OAB according to the definition by the International Continence Society (Haylen et al, 2012) given above.
* Good response to PTNS. For the purpose of this study, responders will be considered those subjects who have achieved a reduction in the number of micturitions per 24 hours by > 30%.
* Able and willing to give informed consent.

Exclusion Criteria:

* Patients who do not comprehend the physiotherapist's instructions or who are unable to co-operate.
* Pregnancy, or plans of becoming pregnant during the course of the study. The main acupuncture point that will be used (SP6) has been reported to induce uterine activity (Hecker et al, 2001).
* Presence of a relevant neurological condition (causing neurogenic detrusor overactivity or peripheral neuropathy).
* Previous history of continence surgery.
* Women with a pace-maker fitted.
* Women with uncorrectable coagulopathies or on anticoagulant medication.
* Presence of dermatological lesions (e.g. dermatitis, eczema...) in the medial aspect of lower leg and/or feet.
* No anticholinergic medication will be allowed during the study period with minimum wash-out period of 15 days before randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Changes in 24-hour micturition frequency | Bladder diaries completed at recruitment and 6 weeks, 12 weeks and 6 months.
  Mean number of micturition episodes recorded in 3-day bladder chart.

SECONDARY OUTCOMES:
Symptom severity | OAB-q completed at recruitment and 6 weeks, 12 weeks and 6 months.
  Severity score on validated OAB-q questionnaire.
Health Related Quality of Life | OAB-q completed at recruitment and 6 weeks, 12 weeks and 6 months.
  HRQoL score as recorded on OAB-q

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Martin-Garcia, MSc, Principal Investigator — Liverpool Women's Hospital
Locations (1):
- Liverpool Women's Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin-Garcia M, Crampton J. A single-blind, randomized controlled trial to evaluate the effectiveness of transcutaneous tibial nerve stimulation (TTNS) in Overactive Bladder symptoms in women responders to percutaneous tibial nerve stimulation (PTNS). Physiotherapy. 2019 Dec;105(4):469-475. doi: 10.1016/j.physio.2018.12.002. Epub 2018 Dec 18. PMID 30862384